CLINICAL TRIAL: NCT07308002
Title: Intermittent (Every-Other-Day) vs Daily Tamsulosin for Men With Lower Urinary Tract Symptoms Secondary to Benign Prostatic Hyperplasia (LUTS/BPH) : A Multicenter, Assessor-Blinded, Randomized Non-Inferiority Trial. Arab Randomized Assessment of BPH Treatment (ARAB Trial)
Brief Title: Intermittent vs Daily Tamsulosin for LUTS/BPH
Acronym: ARAB
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mahmoud Laymon, Prof., Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ARAB BPH Study
Record Dates: First submitted 2025-12-08; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Lower Urinary Tract Symptoms; Prostate Obstruction
Keywords: Lower Urinary Tract Symptoms; Tamsulosin; Benign prostatic obstruction; Alternate-Day Dosing; Ejaculatory Dysfunction
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Ejaculatory Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: After allocation, both investigators and participants will be aware of the assigned dosing regimen (open-label). To minimize bias, all efficacy assessments (e.g., IPSS, uroflowmetry, and PVR) will be conducted by trained assessors who are blinded to treatment allocation and not involved in clinical management or drug dispensing.
  Study statisticians will remain blinded to treatment identity until the database is locked and the primary analysis completed. Any instance of unintentional unblinding will be documented, along with its rationale and potential impact on the study outcome.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Daily arm: Tamsulosin 0.4 mg once daily. (Active Comparator)
  Interventions: Drug: Daily Tamsulosin
- EOD arm: Tamsulosin 0.4 mg every other day (no capsule on off-days) (Experimental)
  Interventions: Drug: Intermittent Tamsulosin

INTERVENTIONS:
Drug: Daily Tamsulosin — Participants receive standard tamsulosin 0.4 mg once daily for the study duration. This arm serves as the reference for evaluating efficacy and safety compared with the intermittent regimen.
  Arms: Daily arm: Tamsulosin 0.4 mg once daily.
Drug: Intermittent Tamsulosin — Participants receive tamsulosin 0.4 mg every other day (intermittent regimen) for the study duration. The regimen is designed to evaluate whether reduced-frequency dosing is non-inferior to standard daily therapy in improving LUTS/BPH symptoms.
  Arms: EOD arm: Tamsulosin 0.4 mg every other day (no capsule on off-days)

SUMMARY:
Background:

Lower urinary tract symptoms (LUTS) are common in aging men, most often due to benign prostatic hyperplasia (BPH), and significantly impair quality of life. α1-adrenoceptor antagonists are first-line therapy, with tamsulosin being the most widely prescribed. However, ejaculatory dysfunction (EjD) is a frequent adverse effect that negatively affects adherence. Optimal dosing strategies that maintain urinary efficacy while reducing EjD are not well defined, and current guidelines provide no recommendations regarding alternate-day dosing.

Patients and Methods:

This multicenter, randomized, open-label, assessor-blinded, parallel-group, non-inferiority trial will enroll men aged ≥50 years with LUTS/BPH and baseline IPSS ≥8. Participants will be randomized 1:1 to receive tamsulosin 0.4 mg once daily or every other day for 24 weeks. The primary endpoint is change in International Prostate Symptom Score (IPSS) from baseline to Week 24. Non-inferiority will be concluded if the upper bound of the two-sided 95% confidence interval (CI) for the between-group difference in mean IPSS change (EOD - Daily) is ≤ +3 points.

The key secondary endpoint is change in Male Sexual Health Questionnaire-Ejaculatory Dysfunction (MSHQ-EjD) total score from baseline to Week 24, tested for superiority only if IPSS non-inferiority is established. Additional secondary endpoints include maximum urinary flow rate (Qmax), post-void residual volume (PVR), IPSS-Quality of Life score, and ejaculatory adverse-event rates.

Sample Size and Analysis:

Assuming an SD of 6 for IPSS change, a non-inferiority margin of +3, one-sided α of 0.025, and 90% power, approximately 85 evaluable patients per arm are required for the primary endpoint. To ensure adequate power for EjD outcomes and allow for 20% attrition, 144 participants per arm (288 total) will be randomized. Analyses will follow the intention-to-treat principle with per-protocol sensitivity analyses. Primary inference will use ANCOVA or MMRM adjusted for baseline score, age, and study site, with multiple imputation for missing data.

Expected Outcomes:

This trial will provide the first adequately powered multicenter evidence on whether every-other-day tamsulosin preserves non-inferior LUTS control while improving ejaculatory outcomes, potentially supporting a simple and cost-effective strategy to enhance tolerability and adherence in men with LUTS/BPH.

DETAILED DESCRIPTION:
Lower urinary tract symptoms (LUTS) due to benign prostatic hyperplasia (BPH) are commonly treated with α1-adrenoceptor antagonists, with tamsulosin being among the most frequently prescribed agents. Although effective for symptom relief, tamsulosin is associated with ejaculatory dysfunction, which may negatively affect treatment satisfaction and adherence. Despite long-standing clinical use, optimal dosing strategies that preserve urinary efficacy while reducing ejaculatory adverse effects remain insufficiently studied. Existing investigations of dose reduction or alternate-day regimens have been limited by small sample size, short follow-up, single-center design, and non-standardized assessment of sexual outcomes. Consequently, international guidelines do not currently recommend every-other-day dosing.

This multicenter, randomized, open-label, assessor-blinded, parallel-group, non-inferiority trial is designed to evaluate whether every-other-day tamsulosin dosing maintains non-inferior improvement in urinary symptoms while offering superior ejaculatory outcomes compared with standard daily dosing. Following a 4-week open-label run-in period with daily tamsulosin, participants demonstrating a predefined clinical response without safety concerns will be randomized in a 1:1 ratio to continue daily dosing or switch to every-other-day dosing for 24 weeks. Randomization will be centralized, computer-generated, and stratified by study site and baseline symptom severity.

After randomization, participants and treating clinicians will be aware of treatment allocation; however, outcome assessors and statisticians will remain blinded to minimize assessment and analytical bias. Study visits and assessments will be standardized across centers, and participants will be instructed not to disclose allocation status to assessors.

Efficacy assessments will include patient-reported symptom scores, objective voiding parameters, and validated sexual function questionnaires collected at prespecified intervals during follow-up. Safety monitoring will include adverse events, orthostatic vital signs, and treatment adherence throughout the study period.

The primary objective is to demonstrate non-inferiority of every-other-day dosing compared with daily dosing for improvement in urinary symptoms over 24 weeks, using a predefined non-inferiority margin based on established clinical relevance. A hierarchical testing strategy will be applied to evaluate superiority for ejaculatory function outcomes only if non-inferiority for urinary symptom control is established. Statistical analyses will follow the intention-to-treat principle with supportive per-protocol analyses, using appropriate regression models adjusted for baseline values and study site.

This study aims to provide high-quality multicenter evidence to inform dosing strategies that optimize both efficacy and tolerability of tamsulosin in men with LUTS/BPH.

ELIGIBILITY:
Inclusion Criteria:

* • Men ≥40 years with LUTS/BPH.

  * IPSS ≥8, Qmax 5-15 mL/s (voided volume ≥150 mL), PVR <200 mL.
  * Sexually active within the past month (for ejaculatory outcomes).
  * BPH-treatment naïve: no prior use of antimuscarinics or 5-α-reductase inhibitors (5-ARIs) and agrees not to initiate these agents during the trial.

Exclusion Criteria:

* • PVR ≥ 200 mL.

  * Prior prostate/ radical pelvic surgery (that affect pelvic innervation).
  * Neurogenic bladder (atonic/ hypotonic bladder).
  * Severe hepatic/renal insufficiency.
  * Significant cardiovascular or cerebrovascular disease.
  * Any indication of surgical treatment (vesical stones, chronic urine retention, recurrent attacks of acute urine retention, recurrent attacks of gross hematuria, hydronephrosis)

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in International prostate symptom score (IPSS) From Baseline to Week 24 | Baseline to Week 24
  Change in the International Prostate Symptom Score (IPSS) from baseline to Week 24. The IPSS is a validated 7-item questionnaire assessing lower urinary tract symptoms, with total scores ranging from 0 to 35, where higher scores indicate more severe symptoms.
  This is a non-inferiority comparison with a non-inferiority margin of +3 IPSS points. Non-inferiority will be concluded if the upper bound of the two-sided 95% confidence interval for the between-group difference in mean IPSS change (Intermittent - Daily) is ≤ +3 points.

SECONDARY OUTCOMES:
Change in MSHQ-Ejaculatory Dysfunction Total Score From Baseline to Week 24 | Baseline to Week 24
  Change in the Male Sexual Health Questionnaire-Ejaculatory Dysfunction (MSHQ-EjD) total score from baseline to Week 24. The MSHQ-EjD is a validated patient-reported outcome measure assessing ejaculatory function, with total scores ranging from 0 to 15, where higher scores indicate better ejaculatory function (less dysfunction).

CONTACTS AND LOCATIONS:
Locations (1):
- Urology and nephrology center, Al Mansurah, Outside U.S./Canada, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Aggregate results will be reported through publications and ClinicalTrials.gov